CLINICAL TRIAL: NCT02778165
Title: My Cardiac Recovery (MyCaRe): A Pilot RCT to Examine the Effect of MyCaRe Android Application on Recovery Outcomes and Enrolment in Cardiac Rehab Post Cardiac Surgery.
Brief Title: My Cardiac Recovery (MyCaRe): A Pilot RCT.
Acronym: MyCaRe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Toronto General Hospital (Other)
Responsible Party: Principal Investigator, Tracey JF Colella, Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-9520
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients receiving usual care are typically referred to CR at the time of discharge from the acute care center via paper or electronic systematic referral (completed by a physician or nurse practitioner). Additionally, a conversation with the patient regarding CR by a healthcare provider may occur, however this communication is not always a consistent occurrence. Once referred, patients will await contact from a CR program in their region/area and if actual program enrollment occurs, this usually happens between 8 to 10 weeks post discharge.
- MyCaRe Android Application (Experimental): The MyCaRe mobile application (education and symptom monitoring which includes pain, mood scales, wound monitoring) and Fitbit accelerometer (steps walked, distance) will be provided to patients receiving intervention group allocation for the initial 6 to 8 weeks recovery post cardiac surgery. The patients will be provided a temporary loan mobile device loaded with MyCaRe and Fitbit Inspire 2 before leaving hospital. They will be asked to input data (pain, mood, wounds, activity, blood sugar, blood pressure) daily if possible in first 2 weeks and once weekly thereafter until 6 to 8 weeks or until entry to a cardiac rehabilitation program.
  Interventions: Other: MyCaRe (my cardiac recovery Android application)

INTERVENTIONS:
Other: MyCaRe (my cardiac recovery Android application) — Android application & Fitbit Inspire 2 activity monitor
  Other Names: MyCaRe
  Arms: MyCaRe Android Application

SUMMARY:
MyCardiacRecovery (MyCaRe) is an interactive platform that includes a standardized educational format and interactive tracking (wound healing and activity progression using photo capabilities and Fitbit Inspire 2 accelerometer) support during the first 6 to 8 weeks post hospital discharge. This android application will help patients and family navigate their way through the continuum of care by providing an: a) integrated link between acute care and outpatient cardiac rehab (CR) for efficient coordination of information and reduction in duplication of services; b) patient care and education materials designed to address salient recovery questions; c) improved communication between the patient and care providers and, d) ensure streamlined systematic referral to CR. This innovative strategy has the potential to positively impact patient satisfaction, improve patient outcomes and possibly minimize financial constraints placed on the health care system. Phase 1 (preliminary usability testing) of prototype 1.0 is complete. Phase 2 will focus on testing MyCaRe 2.0 in a sample of post cardiac surgery patients using a pilot randomized controlled trial (RCT) design.

DETAILED DESCRIPTION:
The early transition period post coronary artery bypass graft surgery is one associated with intense physiological and psychosocial adjustment that requires patients make sustainable long-term lifestyle changes. Cardiac rehabilitation (CR) is an evidence-based risk reduction program that has been shown to improve overall fitness and quality of life as well as lower morbidity and mortality in patients with coronary artery disease. Therefore, the development of supportive strategies to bridge the gap from acute care in to CR through early intervention for cardiac surgery patients is essential. MyCardiacRecovery (MyCaRe) is an interactive platform that includes a standardized educational format and interactive tracking (wound healing and activity progression using photo capabilities and Fitbit Inspire 2 accelerometer) support during the first 6 to 8 weeks post hospital discharge. This application will help patients and family navigate their way through the continuum of care by providing an: a) integrated link between acute care and outpatient cardiac rehab for efficient coordination of information and reduction in duplication of services; b) patient care and education materials designed to address salient recovery questions; c) improved communication between the patient and care providers and, d) ensure streamlined systematic referral to CR. This innovative strategy has the potential to positively impact patient satisfaction, improve patient outcomes and possibly minimize financial constraints placed on the health care system. Phase 1 (preliminary usability testing) of prototype 1.0 is complete. Phase 2 will focus on testing MyCaRe 2.0 in a sample of post cardiac surgery patients using a pilot randomized controlled trial design.

Protocol Summary: App Study Phase 2 - Pilot Randomized Controlled Trial N= 40 (20 usual care + intervention; 20 usual care) Study Population: Post cardiac surgery patient population at 1 acute care cardiac centre in Toronto Study Design Pilot Randomized controlled trial Study Duration March 2022 - Dec 2022 Study Agent/ Intervention MyCaRe prototype (mobile application) Primary Objectives: 1) To examine the effect of MyCaRe application on enrolment in CR post cardiac surgery in comparison to usual care (assessing effectiveness of intervention);

Secondary Objectives:

2) To examine the impact of MyCaRe application on patient recovery and satisfaction (i.e. knowledge level, perceptions of recovery outcomes such as activity progression, quality of life, anxiety and depression) 3) To examine the effect of MyCaRe application on health services use. 4) To examine patient and clinician satisfaction, specifically user ease, usability and comfort with MyCaRe application.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the sample includes:

1. comprehend/understand instructions for study and use of app/Fitbit,
2. > 35 years of age,
3. undergoing traditional (sternotomy approach) coronary artery bypass graft (CABG) surgery,
4. an uncomplicated postoperative course,
5. standard length of hospital stay (four to eight days),
6. access to wifi internet in their home,
7. able to hear telephone conversation,
8. reside within the greater Toronto region (GTA) or if outside GTA willing to return devices via mail upon completion of study.

Exclusion Criteria:

* The exclusion criteria will include those persons who:

  1. have cardiac surgery procedures other than CABG,
  2. reside in a nursing home or long term care facility,
  3. have any neurological or psychiatric disorder that may impede their ability to self reflect or communicate,
  4. sustained in-hospital post surgical complications of major significance (such as stroke, deep wound infections, pericardial effusion, etc.), 5) inability to ambulate (i.e. walk unaided at 2 mph).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Enrolment in cardiac rehabilitation | 8 weeks post operative discharge
  The number of individuals who attend their initial cardiac rehab intake appointment will be the primary outcome measure of enrollment. Enrollment is defined in accordance with Canadian Cardiovascular Society data definitions (http://bridge.ccs.ca/index.php/en/), as patient having attended their scheduled cardiac rehab intake appointment (i.e., risk factor assessment, goal-setting). Enrollment will be verified with patient as well as with the CR program in which they are enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey J Colella, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Cardiac Rehabilitation, Rumsey Centre, TRI-UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardiac Care Network of Ontario. Report on adult cardiac surgery in Ontario. Retrieved July 2, 2013 at http://www.ccn.ca/ccc public/uploadfiles/files/Provincial%21 Cardiac%20Surgery%20Reports%20-%20Final%20Draft.pdf
- [Background] Stewart, M.J. (1993). Integrating social support in nursing. Newbury Park: Sage.
- [Background] Goodman H. Patients' perceptions of their education needs in the first six weeks following discharge after cardiac surgery. J Adv Nurs. 1997 Jun;25(6):1241-51. doi: 10.1046/j.1365-2648.1997.19970251241.x. PMID 9181423
- [Background] Meleis AI. Transition Theory. Middle range and situation specific theories in nursingresearch and practice. 2010. Springer Publishing: New York.
- [Background] Hamalainen H, Smith R, Puukka P, Lind J, Kallio V, Kuttila K, Ronnemaa T. Social support and physical and psychological recovery one year after myocardial infarction or coronary artery bypass surgery. Scand J Public Health. 2000 Mar;28(1):62-70. doi: 10.1177/140349480002800111. PMID 10817316
- [Background] Lapum J, Angus JE, Peter E, Watt-Watson J. Patients' discharge experiences: returning home after open-heart surgery. Heart Lung. 2011 May-Jun;40(3):226-35. doi: 10.1016/j.hrtlng.2010.01.001. Epub 2010 Apr 14. PMID 20561868
- [Background] World Health Organization (WHO). 2005 Facing the facts: The impact of chronic disease in Canada. Retrieved May 4, 2011 at http://www.who.int/chp/chronic_disease_report/en/
- [Background] Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP; Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Secondary prevention through cardiac rehabilitation: from knowledge to implementation. A position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur J Cardiovasc Prev Rehabil. 2010 Feb;17(1):1-17. doi: 10.1097/HJR.0b013e3283313592. PMID 19952757
- [Background] Alter DA, Oh PI, Chong A. Relationship between cardiac rehabilitation and survival after acute cardiac hospitalization within a universal health care system. Eur J Cardiovasc Prev Rehabil. 2009 Feb;16(1):102-13. doi: 10.1097/HJR.0b013e328325d662. PMID 19165089
- [Background] Arthur HM, Suskin N, Bayley M, Fortin M, Howlett J, Heckman G, Lewanczuk R. The Canadian Heart Health Strategy and Action Plan: Cardiac rehabilitation as an exemplar of chronic disease management. Can J Cardiol. 2010 Jan;26(1):37-41. doi: 10.1016/s0828-282x(10)70336-6. PMID 20101356
- [Background] Oldridge N. Exercise-based cardiac rehabilitation in patients with coronary heart disease: meta-analysis outcomes revisited. Future Cardiol. 2012 Sep;8(5):729-51. doi: 10.2217/fca.12.34. PMID 23013125
- [Background] Taylor RS, Brown A, Ebrahim S, Jolliffe J, Noorani H, Rees K, Skidmore B, Stone JA, Thompson DR, Oldridge N. Exercise-based rehabilitation for patients with coronary heart disease: systematic review and meta-analysis of randomized controlled trials. Am J Med. 2004 May 15;116(10):682-92. doi: 10.1016/j.amjmed.2004.01.009. PMID 15121495
- [Background] Li J, Siegrist J. Physical activity and risk of cardiovascular disease--a meta-analysis of prospective cohort studies. Int J Environ Res Public Health. 2012 Feb;9(2):391-407. doi: 10.3390/ijerph9020391. Epub 2012 Jan 26. PMID 22470299
- [Background] Schuler G, Adams V, Goto Y. Role of exercise in the prevention of cardiovascular disease: results, mechanisms, and new perspectives. Eur Heart J. 2013 Jun;34(24):1790-9. doi: 10.1093/eurheartj/eht111. Epub 2013 Apr 7. PMID 23569199
- [Background] Jackson L, Leclerc J, Erskine Y, Linden W. Getting the most out of cardiac rehabilitation: a review of referral and adherence predictors. Heart. 2005 Jan;91(1):10-4. doi: 10.1136/hrt.2004.045559. PMID 15604322
- [Background] Colella TJ, Gravely S, Marzolini S, Grace SL, Francis JA, Oh P, Scott LB. Sex bias in referral of women to outpatient cardiac rehabilitation? A meta-analysis. Eur J Prev Cardiol. 2015 Apr;22(4):423-41. doi: 10.1177/2047487314520783. Epub 2014 Jan 28. PMID 24474091
- [Background] Cook D, et al. (Discovery Project). Mayo Clinic pilots myCare iPad app for cardiac surgery support, engaging patients & families. Feb, 5, 2013; Retrieved from: http://consumerehealthengagement.squarespace.com/consumerehealthengagement/2013/2/5/mayo-pilots-mycare-ipad-app-for-cardiac-surgery-support-enga.html
- [Background] Seto E, Leonard KJ, Cafazzo JA, Barnsley J, Masino C, Ross HJ. Mobile phone-based telemonitoring for heart failure management: a randomized controlled trial. J Med Internet Res. 2012 Feb 16;14(1):e31. doi: 10.2196/jmir.1909. PMID 22356799
- [Background] Hirano, SH, Tang KP, Cheng KG, Hayes GR. The Estrellita system: A health informatics tools to support caregivers of preterm infants 2012; doi 10.4108/cst.pervasivehealth.2012.248718
- [Background] Sieverdes JC, Treiber F, Jenkins C, Hermayer K. Improving diabetes management with mobile health technology. Am J Med Sci. 2013 Apr;345(4):289-295. doi: 10.1097/MAJ.0b013e3182896cee. PMID 23531961
- [Background] Maddison R, Whittaker R, Stewart R, Kerr A, Jiang Y, Kira G, Carter KH, Pfaeffli L. HEART: heart exercise and remote technologies: a randomized controlled trial study protocol. BMC Cardiovasc Disord. 2011 May 31;11:26. doi: 10.1186/1471-2261-11-26. PMID 21624142
- [Background] Ritchie C, Richman J, Sobko H, Bodner E, Phillips B, Houston T. The E-coach transition support computer telephony implementation study: protocol of a randomized trial. Contemp Clin Trials. 2012 Nov;33(6):1172-9. doi: 10.1016/j.cct.2012.08.007. Epub 2012 Aug 19. PMID 22922245
- [Background] Reid RD, Morrin LI, Beaton LJ, Papadakis S, Kocourek J, McDonnell L, Slovinec D'Angelo ME, Tulloch H, Suskin N, Unsworth K, Blanchard C, Pipe AL. Randomized trial of an internet-based computer-tailored expert system for physical activity in patients with heart disease. Eur J Prev Cardiol. 2012 Dec;19(6):1357-64. doi: 10.1177/1741826711422988. Epub 2011 Sep 8. PMID 21903744
- [Background] . Liu J. Seamless Mobile Health. 2012. Retrieved May 28, 2013 from www.seamlessmobilehealth.ca
- [Background] Lawson, Telus Health, Canada Health Infoway and Mental Health Engagement Network retrieved on July 2, 2013 at http://www.telushealth.com/news-and-events/news-releases/release/2012/10/12/lawson-telus-health-and-canada-health-infoway-launch-the-mental-health-engagement-network-initiative-to-measure-effectiveness-of-new-technology-in-ongoing-health-management
- [Background] Topol, E. The creative destruction of medicine: How the digital revolution will create better health care, 2012; Basic, New York.
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Artinian NT, Duggan CH. Sex differences in patient recovery patterns after coronary artery bypass surgery. Heart Lung. 1995 Nov-Dec;24(6):483-94. doi: 10.1016/s0147-9563(95)80026-3. PMID 8582824
- [Background] Chunta KS. Expectations, anxiety, depression, and physical health status as predictors of recovery in open-heart surgery patients. J Cardiovasc Nurs. 2009 Nov-Dec;24(6):454-64. doi: 10.1097/JCN.0b013e3181ac8a3c. PMID 19858954
- [Background] Bandura, A. (1986). Social foundation of thought and action: A social cognitive theory. Englewood Cliffs, NJ: Prentice-Hall.
- [Background] Cohen, S., Underwood, L.G. & Gottlieb, B.H. (2000). Social support measurement and intervention: A guide for health and social scientists. New York: Oxford University Press
- [Background] Parent N, Fortin F. A randomized, controlled trial of vicarious experience through peer support for male first-time cardiac surgery patients: impact on anxiety, self-efficacy expectation, and self-reported activity. Heart Lung. 2000 Nov-Dec;29(6):389-400. doi: 10.1067/mhl.2000.110626. PMID 11080319
- [Background] Dafoe W, Arthur H, Stokes H, Morrin L, Beaton L; Canadian Cardiovascular Society Access to Care Working Group on Cardiac Rehabilitation. Universal access: but when? Treating the right patient at the right time: access to cardiac rehabilitation. Can J Cardiol. 2006 Sep;22(11):905-11. doi: 10.1016/s0828-282x(06)70309-9. PMID 16971975
- [Background] Gortner S.R., Jaeger A.A., Harr J., & Hlatky M.A. Elders' recovery from cardiac surgery: Is gender a factor? Journal of Myocardial Ischemia, 1994; 6(9), 17-25.
- [Background] King KM, Gortner SR. Women's short-term recovery from cardiac surgery. Prog Cardiovasc Nurs. 1996 Spring;11(2):5-15. PMID 8718958
- [Background] King KM. Gender and short-term recovery from cardiac surgery. Nurs Res. 2000 Jan-Feb;49(1):29-36. doi: 10.1097/00006199-200001000-00005. PMID 10667626
- [Background] Grace SL, Chessex C, Arthur H, Chan S, Cyr C, Dafoe W, Juneau M, Oh P, Suskin N. Systematizing Inpatient Referral to Cardiac Rehabilitation 2010: Canadian association of cardiac rehabilitation and Canadian cardiovascular society joint position paper. J Cardiopulm Rehabil Prev. 2011 May-Jun;31(3):E1-8. doi: 10.1097/HCR.0b013e318219721f. PMID 21460733
- [Background] Takacs J, Pollock CL, Guenther JR, Bahar M, Napier C, Hunt MA. Validation of the Fitbit One activity monitor device during treadmill walking. J Sci Med Sport. 2014 Sep;17(5):496-500. doi: 10.1016/j.jsams.2013.10.241. Epub 2013 Oct 31. PMID 24268570
- [Background] Giannakidou DM, Kambas A, Ageloussis N, Fatouros I, Christoforidis C, Venetsanou F, Douroudos I, Taxildaris K. The validity of two Omron pedometers during treadmill walking is speed dependent. Eur J Appl Physiol. 2012 Jan;112(1):49-57. doi: 10.1007/s00421-011-1951-y. Epub 2011 Apr 9. PMID 21479653
- [Background] Mitchell PH, Powell L, Blumenthal J, Norten J, Ironson G, Pitula CR, Froelicher ES, Czajkowski S, Youngblood M, Huber M, Berkman LF. A short social support measure for patients recovering from myocardial infarction: the ENRICHD Social Support Inventory. J Cardiopulm Rehabil. 2003 Nov-Dec;23(6):398-403. doi: 10.1097/00008483-200311000-00001. No abstract available. PMID 14646785
- [Background] Berkman LF, Blumenthal J, Burg M, Carney RM, Catellier D, Cowan MJ, Czajkowski SM, DeBusk R, Hosking J, Jaffe A, Kaufmann PG, Mitchell P, Norman J, Powell LH, Raczynski JM, Schneiderman N; Enhancing Recovery in Coronary Heart Disease Patients Investigators (ENRICHD). Effects of treating depression and low perceived social support on clinical events after myocardial infarction: the Enhancing Recovery in Coronary Heart Disease Patients (ENRICHD) Randomized Trial. JAMA. 2003 Jun 18;289(23):3106-16. doi: 10.1001/jama.289.23.3106. PMID 12813116
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Freund T, Gensichen J, Goetz K, Szecsenyi J, Mahler C. Evaluating self-efficacy for managing chronic disease: psychometric properties of the six-item Self-Efficacy Scale in Germany. J Eval Clin Pract. 2013 Feb;19(1):39-43. doi: 10.1111/j.1365-2753.2011.01764.x. Epub 2011 Aug 23. PMID 21883720
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Whelan-Goodinson R, Ponsford J, Schonberger M. Validity of the Hospital Anxiety and Depression Scale to assess depression and anxiety following traumatic brain injury as compared with the Structured Clinical Interview for DSM-IV. J Affect Disord. 2009 Apr;114(1-3):94-102. doi: 10.1016/j.jad.2008.06.007. Epub 2008 Jul 25. PMID 18656266
- [Background] Dempster M, Donnelly M, Fitzsimmon D. Generic, disease-specific and individualized approaches to measuring health -related quality of life among people with heart disease - a comparative analysis. Psychology & Health. 2002 ;17 ;447-457.
- [Background] Gardner JK, McConnell TR, Klinger TA, Herman CP, Hauck CA, Laubach CA Jr. Quality of life and self-efficacy: gender and diagnoses considerations for management during cardiac rehabilitation. J Cardiopulm Rehabil. 2003 Jul-Aug;23(4):299-306. doi: 10.1097/00008483-200307000-00007. PMID 12894004
- [Background] McConnell TR, Laubach CA, Memon M, Gardner JK, Klinger TA, Palm RJ. Quality of Life and Self Efficacy in Cardiac Rehabilitation Patients Over 70 Years of Age Following Acute Myocardial Infarction and Bypass Revascularization Surgery. Am J Geriatr Cardiol. 2000 Jul;9(4):210-218. doi: 10.1111/j.1076-7460.2000.80040.x. PMID 11416568
- [Background] Colella TJF, King KM. The effect of a professionally-guided telephone peer support intervention on early recovery outcomes in men following coronary artery bypass graft surgery. Doctoral dissertation University of Calgary, CAN. Under review Soc Sci Med, 2016.
- [Background] Shanmugasegaram S, Gagliese L, Oh P, Stewart DE, Brister SJ, Chan V, Grace SL. Psychometric validation of the cardiac rehabilitation barriers scale. Clin Rehabil. 2012 Feb;26(2):152-64. doi: 10.1177/0269215511410579. Epub 2011 Sep 21. PMID 21937522
- [Background] Grace SL, Shanmugasegaram S, Gravely-Witte S, Brual J, Suskin N, Stewart DE. Barriers to cardiac rehabilitation: DOES AGE MAKE A DIFFERENCE? J Cardiopulm Rehabil Prev. 2009 May-Jun;29(3):183-7. doi: 10.1097/HCR.0b013e3181a3333c. PMID 19471138
- [Background] Grace SL, Gravely-Witte S, Kayaniyil S, Brual J, Suskin N, Stewart DE. A multisite examination of sex differences in cardiac rehabilitation barriers by participation status. J Womens Health (Larchmt). 2009 Feb;18(2):209-16. doi: 10.1089/jwh.2007.0753. PMID 19183092
- [Background] Brooke J. The system usability scale. http://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html
- [Result] Kmill C, Sherrington L, Third G. Increasing access to cardiac rehabilitation through telemedicine technology. Can Nurse. 2007 May;103(5):8-9. No abstract available. PMID 17555156
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536